CLINICAL TRIAL: NCT04968067
Title: Effectiveness of the Professional-led Support Programme Using a Mobile Application Versus Phone Advice on Patients at Risk of Coronary Heart Disease - A Randomized Controlled Trial (Phase 2)
Brief Title: A Programme Using a Mobile Application Versus Phone Advice on Patients at Risk of Coronary Heart Disease - A RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Tung Wah College (Other)
Responsible Party: Principal Investigator, Dr Eliza Wong, Principal investigator, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HSEARS20201218002
Record Dates: First submitted 2021-07-13; First posted 2021-07-20 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Coronary Heart Disease
Keywords: e-health; nursing telephone advice; exercise; risk factors
MeSH Terms: conditions — Coronary Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study will employ a prospective randomized controlled trial (RCT) with two arms, namely, the App group, NTA (nursing telephone advice) group. This design is guided by the CONSORT checklist
Who Masked: Investigator, Outcomes Assessor
Masking Description: To minimize subject contamination, the different groups will be assigned different follow-up dates. The research assistants who are responsible for collecting data will be blinded to the group allocations. To ensure allocation concealment, each computer generated sequence will be put in a sequentially numbered, opaque sealed envelope. The envelope will be opened by RA1 after the participant has completed the baseline questionnaire.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App group (Experimental): In addition to the usual care, the participant will receive a health talk , a CHD app and a briefing from a trained research nurse (A). The app provides features such as structured e-educational contents and supportive features such as knowledge platform and member area.
  Interventions: Device: App group
- Nursing telephone advice (NTA) group (Active Comparator): In addition to the above usual care, the participant will receive a health talk , three monthly 20-minute telephone follow-ups supplemented by take home leaflet will be provided by a trained research nurse for up to 3 months. Patients can ask about their related health problems, if any. The team has set up a telephone advice guide to support the research nurse in giving phone advice and text messages.
  Interventions: Device: Nursing telephone advice (NTA) group

INTERVENTIONS:
Device: App group — In addition to the usual care, the participant will receive a health talk related to CHD care, a CHD app and a briefing from a trained research nurse (A). The app provides features such as structured e-educational contents and supportive features such as knowledge platform and member area.
  Arms: App group
Device: Nursing telephone advice (NTA) group — All subjects will continue their usual care with prescribed medical treatments and follow-ups if any. By appointment, a trained nurse will provide a health talk related to the CHD care. In addition to the above usual care, three monthly 20-minute telephone follow-ups supplemented by take home leaflet will be provided by a trained research nurse for up to 3 months. Patients can ask about their related health problems, if any. The team has set up a telephone advice guide to support the research nurse in giving phone advice and text messages. .In summary, all two groups will receive from a nurse similar educational content as that related to their CHD and care. The only difference will be the re-enforcement and continual support provided through an app, telephone nursing advice and leaflet.
  Arms: Nursing telephone advice (NTA) group

SUMMARY:
It aims to compare the effects of a professional -led support programme using a mobile application versus telephone advice on clients at risk of coronary heart disease. A multi-centre, single-blinded, randomized controlled trial will be conducted. 168 Clients who are at risk of coronary heart disease (CHD), able to use a smart phone will be randomized into the App Support group (App group) or the Nursing Telephone advice (NTA) group . All participants will receive same nursing educational briefing related to CHD. The App Group will additional receive an app use to support their self care whereas the NTA group will receive nursing telephone advice for 20 minutes monthly.

Health outcomes will be collected at baseline (T0), 1 months (T1), 3 months (T2). Data analysis will be conducted using a Generalized Estimating Equations model to assess differential changes in all outcome variables.

DETAILED DESCRIPTION:
The aim of this study is to test the effects of a professional-led support programme for clients who are at risk of developing CHD on outcomes of total exercise, self-efficacy and self-management behavior, emergency department attendance and hospitalizations, CHD risk factor profile, and quality of life.

Over 3 months, the investigators will examine the effect on the App group as compared to the NTA group and the control group of: Total amount of exercise (primary outcome) and secondary outcomes:1) Self-efficacy and self-management behavior; 2)Emergency department attendance and hospitalization frequency;3) CHD risk factor profile (smoking, blood pressure, body mass index, blood lipid level);4) Cardiovascular functional endurance;5)Perceived stress ; and 6) Quality of life.

A prospective multi-Centre, parallel, randomized controlled trial (RCT) with two arms - an app support programme (App) group vs a Nursing Telephone advice (NTA) group and a control group - will be adopted. The RCT method follow CONSORT 2010 guideline. 168 subjects will be required (n=84 each group). Subject recruitment will likely take about 14 months.

Intervention protocol: 168 Clients who are at risk of coronary heart disease (CHD), able to use a smart phone will be randomized into the App Support group (App group) or the Nursing Telephone advice (NTA) group. All eligible participants will receive same nursing educational briefing related to CHD. The App Group will additionally receive an app use to support their self -care whereas the NTA group will receive a leaflet and a monthly nursing telephone advice ( about 20 minutes per call. The duration of intervention will be about 3 months. Health outcomes will be collected by research assistant at baseline (T0), 1 months (T1), 3 months (T2) at the community Centre or research Centre. Data analysis will be conducted using SPSS and a Generalized Estimating Equations model to assess differential changes in all outcome variables. All the tests will be two-sided and a p-value of <0.05 will be considered statistically significant.

Ethical approval and permission will be sought from the study university and the selected community centres. RCT registration has been obtained from the ClinicalTrials.gov Protocol Registration system (https://clinicaltrials.gov/).

ELIGIBILITY:
The study's subject inclusion criteria will be:

1. Chinese adults with coronary cardiac risk factors (at least two from iv );
2. those able to perform a brisk walking exercise; and
3. those who possess a smart phone and are able to use it.
4. Coronary heart disease risk factors:

   * current regular smoker,
   * over 50 years of age;
   * has a medical diagnosis of diabetes or hypertension;
   * has a family history of ischaemic heart disease or hyperlipaemia ;
   * has hyperlipidaemia or is regularly taking drugs for hyperlipidaemia;
   * is obese (BMI>25);
   * has had a Percutaneous Coronary Intervention performed;
   * was diagnosed with stable angina and prescribed with Trinitroglycerin (TNG) drugs.

The exclusion criteria will be those :

1. with mental, visual, hearing, or cognitive impairments as a result of which they are unable to perform a brisk walking exercise or communicate using a smart phone;
2. on a waiting list for cardiac angiography within 6 months, and
3. has medical diagnosis of unstable angina.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-10-30 (Estimated); Study Completion 2023-06-03 (Estimated)

PRIMARY OUTCOMES:
Change of total physical exercise: the Godin-Shepherd Leisure Time Physical Activity Questionnaire. | baseline, 3 months
  This scale measures the frequency, duration the respondent has performed strenuous, moderate and mild exercise outside of their work duties. The total weekly leisure activity is calculated in arbitrary units as a sum of the products of the separate components

SECONDARY OUTCOMES:
Change of Self-efficacy in illness management | baseline, 3 months
  Six items of Self-efficacy in illness management from The Chinese Self-Management Behaviour Questionnaire was used. It was originally developed by Lorig, and the Chinese language version was translated and validated by Siu et al. in Hong Kong. A final subtotal sum of score could be calculated to assess their self efficacy level.
Change of blood pressure | baseline, 3 months
  systolic and distolic pressure will be collected by research assistant
Change of cardiovascular endurance test | baseline, 3 months
  Three-minute step test aims to test the client's cardiovascular functional endurance after exercise across the age span and gender. A participant step on and off of a 12-inch high bench/ or stair for 3 minutes. Their pulse is then taken while the participant remains standing. Compare the heart rate with the table according to the age and gender to determine the fitness within a range of 7 scores from excellent to good, above average, average, below average, poor and very poor.
Change of total physical exercise | baseline, 3 months
  This outcome will be measured using the Godin-Shepherd Leisure Time Physical Activity Questionnaire. This scale measures how often per week and how long per session the respondent has performed strenuous, moderate and mild exercise outside of their work duties.
Change of perceived stress scale (PSS-10) | baseline, 3 months
  10 self-reported items are used to measure the degree to which situation in a person's life are considered stressful, as well as the current levels of stress experienced in the last month. The summative scores range from 0 to 40, with higher scores indicating higher stress levels. These scores have been used previously to assess the experienced level of stress as an outcome measure and have good psychometric properties in cardiac patients.
Change of Quality of Life:ED-5D | baseline, 3 months
  The ED-5D is a generic instrument used to measure the quality of life in patients with cardiovascular disease in Chinese and other populations. These scale is divided into 5 parts: mobility, self-care, usual activities, pain/discomfort and anxiety/ depression. Participants are asked to respond to the items using the following options: no problem, moderate problems, and extreme problems. The 5 items will also be ranked on a visual analogue scale (VAS) with a range with points from 0 (worst possible health) to 100 (best possible health) to assess the patient's health. The ED-5D was found to be satisfactorily valid and reliable in many populations, including CHD patients.
Hospitalization frequency | 3 months
  frequency of hospitalization will be asked.
change of body weight | baseline, 3 months
  body weight will be measured by RA
change in LDL cholesterol | baseline, 3 months
  Blood samples for measuring LDL cholesterol will be taken by using a finger stick using auto-analysed and the participants are asked to have 8 hours fasting.
Change in HDL cholestero | baseline, 3 months
  Blood samples for measuring HDL cholesterol will be taken by using a finger stick using auto-analysed and the participants are asked to have 8 hours fasting.

CONTACTS AND LOCATIONS:
Overall Officials: Eliza ML wong, PhD, Principal Investigator — Tung Wah College
Locations (1):
- Wan chai Methodist Centre for the Seniors, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No